CLINICAL TRIAL: NCT06199947
Title: Study of the Role of Oncostatin M in Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROMCOR
Record Dates: First submitted 2023-11-14; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer; Cytokine
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Samples (Experimental)
  Interventions: Other: Biopsies and Blood collection

INTERVENTIONS:
Other: Biopsies and Blood collection — Each participant will have 2 additionnal biopsies during his/her diagnostic endoscopy plus two blood test during his/her inclusion

SUMMARY:
The ROMCOR study will be interested in the impact and the role of oncostatin M (OSM), a cytokine belonging to IL-6 superfamily, in the physiopathology of head and neck squamous cell carcinoma. The study team will study the impact of the presence of OSM and its main receptor OSM-R2 on several survival outcomes (overall survival, progression free survival) by multiple technics such as immunohistochemistry, transcriptomic in situ assays and spatial transcriptomic. Furthermore, the study team will try to show a link between serum level of several cytokines and in situ tumoral OSM.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age;
* with suspected squamous cell carcinoma of the oral cavity, oropharynx or pharyngolarynx (any stage);
* with healthy, untreated contralateral mucosa and no contraindications to biopsy;
* with no history of any type of cancer;
* with a WHO performance status index of 0 to 2 inclusive ;
* able to receive treatment according to current European Society of Medical Oncology guidelines ;
* without guardianship, curatorship or subordination;
* benefiting from a Social Security scheme or benefiting from one through a third party;
* have given informed consent to participate in the study.

Exclusion Criteria:

* previously pre-treated in the ear, nose, throat sphere by radiotherapy or having already received anti-cancer chemotherapy;
* on long-term immunosuppressive therapy, defined as taking an immunosuppresseur, identified as such in the ATC classification, for 7 days, cortico-therapy > 7.5mg/day for more than 3 months, treatment or history of anti-CD20 treatment within the year, or regular plasmatic exchange or gamma globulin infusion;
* benefiting from enhanced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection;
* pregnant or breast-feeding women of childbearing age (menopause must be documented and more than 2 years old) who refuse or do not have an effective method of contraception (hormonal/mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy) for the duration of the study.
* final diagnosis of non-squamous cell carcinoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To analyze the relative expression of OSM, several inflammatory cytokines and their receptors in head and neck squamous cell carcinomas (SCC). | 1 month
  The relative expression of transcripts for OSM, OSM-R, as well as the main inflammatory cytokines and their receptors (LIFR, Gp130, IL-31, IL6, IL-1β, TNF-α, IL-4, IL-10, IL-34, CXCL8, CXCL2, IL-17 and GCSF) will be compared between tumor and non-tumor biopsy samples.
  These comparisons will also be stratified by disease stage (localized, locally advanced, metastatic).
  Cytokine expression will be studied by RT-qPCR after RNA extraction and retro-transcription on frozen tissue biopsies (tumor and non-tumor) in nitrogen, and the value will be expressed in relation to the expression of two common housekeeping genes, GADPH and Actin B.

SECONDARY OUTCOMES:
Analysis of the tumor immune cell microenvironment that secret OSM in head and neck squamous cell carcinoma with the cell-selectine RNA sequencing method. | 1 month
  To know what type of cells secrete OSM in the microenvironment, we will use GeoMx Nanostring (c) technique. It consists of a selective RNA or protein sequecing of immunofluorescence labelled cells on parrafine embedded tissues. Investigators will then label OSM-secreting cells with anti-OSM fluorochrome and collect it to be sequenced
Relative expression by RT-qPCR of epithelial-mesenchymal transition (EMT) transcripts will be compared in tumoral mucosa versus normal mucosa of patients | 1 month
  Investigators will study the following genes : SNAI1, SERPIN B3, TGM2, ZEB1, YAP-1, FAT-1, CK13, VIM, OCT-4, SOX-2, CD-44, BMI-1 and KLF-4
Correlation between relative expression of OSM and OSM-R by RT-qPCR and the relative expression of epithelial-mesenchymal transition transcripts in tumoral mucosa | 1 month
  Investigators will study the following genes : SNAI1, SERPIN B3, TGM2, ZEB1, YAP-1, FAT-1, CK13, VIM, OCT-4, SOX-2, CD-44, BMI-1 and KLF-4
Caracterisation of the prognostic impact of tissue-level immunohistochemistry expression of OSM and OSM-R at diagnosis on progression-free survival. | 18 month
  Tissues will be classified as OSM positive (positive staining) or negative (no staining) and OSM-R positive or negative. Progression-free survival of positive and negative patients will be compared.
  PFS will be defined as a composite criterion :progression of the mesurable target > 20%, progression > 20% AND at least 5mm and emergence of new lesions PFS will be mesured at 12 and 18 months
Caracterisation of the prognostic impact of transcriptomic expression of OSM and OSM-R at diagnosis on progression-free survival. | 18 month
  Biopsies will be classified as OSM / OSM-R overexpressing tissue (ratio : relative expression of OSM and OSM-R in tumoral mucosa / relative expression of OSM and OSM-R in normal mucosa by RT-qPCR is above the median) or underexpressing tissue (ratio under the median).
  Progression-free survival of overexpressing and underexpressing patients will be compared.
  PFS will be defined as a composite criterion :progression of the mesurable target > 20%, progression > 20% AND at least 5mm and emergence of new lesions PFS will be mesured at 12 and 18 months
Correlation between serum concentrations of OSM and several circulating inflammatory cytokines and their respective expression in tumor tissue in head and neck squamous cell carcinoma at diagnosis. | 1 month
  OSM and other cytokines (LIFR, le Gp130, l'IL-31, l'IL6, l'IL-1β, le TNF-α, l'IL-4, l'IL-10, l'IL-34, le CXCL8, le CXCL2, l'IL-17 et le GCSF) will be analysed by the semi-quantitative ELISA technique on patients's sera.
  Same cytokines will be assessed in tumoral mucosa by RT-qPCR. Comparison between their relative expression by RT-qPCR and their serum concentration will be study
Caracterisation of the prognostic impact of serum OSM concentrations at diagnosis on progression-free survival | 1 month
  Patients will be classified as high serum concentration of OSM at baseline or low serum concentration at baseline (concentration cut-off not known in literature) using the semi-quantitative ELISA technique.
  Progression-free survival of overexpressing and underexpressing patients will be compared.
  PFS will be defined as a composite criterion :progression of the mesurable target > 20%, progression > 20% AND at least 5mm and emergence of new lesions PFS will be mesured at 12 and 18 months
Caracterisation of the relationship between changes in serum cytokine concentrations (between the time of diagnosis and 3 months after the end of initial treatment) and early response to treatment (3 months after the end of initial treatment). | 18 month
  For each cytokines dosed in serum, we will describe if the variation of their concentrations (R= T0 - (T0+Dt/T0))*100 ) as an impact on the response at 3 month (defined as the V2 visit).
  Reponse rate is defined as (RECIST v1.1) :
  complete response : no residual disease is clinically or radiologically assessable at 3 month partial response : decrease of the mesurable targets of more than 30% but still assessable stable disease : modification of the mesurable targets between a decrease of less than 30% and a progression of less than 20% progression : progression of the mesurable targets of more than 20%